CLINICAL TRIAL: NCT02683148
Title: A Phase I/II Clinical Trial of Dose-Escalating DHEA in Synovial Sarcoma Patients
Brief Title: DHEA in Synovial Sarcoma Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial did not show any positive effects.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201603100
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Synovial Sarcoma; Sarcoma, Synovial
MeSH Terms: conditions — Sarcoma, Synovial | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: DHEA Dose Level 1 (Experimental): -DHEA is an oral supplement which will be administered on an outpatient basis at the prescribed dose daily on a 28-day cycle.
  Interventions: Drug: DHEA; Other: FACT-67 validated survey
- Arm 2: DHEA Dose Level 2 (Experimental): -DHEA is an oral supplement which will be administered on an outpatient basis at the prescribed dose daily on a 28-day cycle.
  Interventions: Drug: DHEA; Other: FACT-67 validated survey
- Arm 3: DHEA Dose Level 3 (Experimental): -DHEA is an oral supplement which will be administered on an outpatient basis at the prescribed dose daily on a 28-day cycle.
  Interventions: Drug: DHEA; Other: FACT-67 validated survey
- Arm 4: DHEA Phase II (Experimental): -DHEA is an oral supplement which will be administered on an outpatient basis at the prescribed dose daily on a 28-day cycle.
  Interventions: Drug: DHEA; Other: FACT-67 validated survey

INTERVENTIONS:
Drug: DHEA
  Other Names: Dehydroepiandrosterone
Other: FACT-67 validated survey — * Baseline, Cycle 1 Day 15, and Day 1 of each cycle beginning with Cycle 2
  * 7 questions with answers ranging from 0=Not At All to 4 = Very Much.

SUMMARY:
DHEA is a natural allosteric inhibitor of glucose-6-phosphate dehydrogenase (G6PD). G6PD is a key regulatory enzyme for the survival of synovial sarcoma. The investigators postulate that they can inhibit the production of NADPH in synovial sarcoma and cause cell death by using a naturally occurring G6PD inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed metastatic or non-resectable synovial sarcoma.
* Failed at least one line of chemotherapy. Neoadjuvant and adjuvant chemotherapy count as a prior line of therapy.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* At least 16 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 50,000/mcl
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Patients using antiestrogens for oral birth control are ineligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* A history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to DHEA or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with DHEA. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Known mania-associated psychiatric disorder.
* Known seizure disorder.
* Using corticosteroids or estrogen-based oral birth control.
* Using drugs known to lower or increase levels of DHEA.
* Requires estrogen or testosterone.
* Taking warfarin sodium. Patients on other blood thinners should be monitored for thrombocytopenia.
* Taking a strong inhibitor or inducer of cytochrome P450. Intermediate inhibitors are allowed if deemed medically necessary.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of DHEA (Phase I only) | Completion of cycle 1 for all phase I patients (estimated to be 2 years)
  * MTD is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose escalations will proceed until the MTD has been reached.
  * Dose-limiting toxicities are defined as one of the following events occurring during the 1st cycle of treatment thought to be possibly, probably, or definitely related to treatment:
    * Grade 3 or greater liver function test abnormalities
    * Grade 3 or greater psychiatric disorder
    * Quality of life (QOL) alteration (change in score of 30%)
Progression-free rate (complete response + partial response + stable disease) (Phase II only) | Up to 5 years
  * Complete response (CR): disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) must have reduction inf short axis to <10mm, disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial response (PR): at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diaters while on study

SECONDARY OUTCOMES:
Rate of progression-free survival (PFS) (Phase II only) | 3 months
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease (PD): aAppearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Toxicity of DHEA as measured by grade and frequency of adverse events | 30 days after completion of treatment (estimated to be 7 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Van Tine, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu